CLINICAL TRIAL: NCT07009301
Title: An Observational Study About a Case of Pulmonary Embolism Following Viper's Bite
Brief Title: Pulmonary Embolism Following Viper's Bites: A Case Report
Status: Completed | Type: Observational
Sponsor: Younes Oujidi (Other)
Responsible Party: Sponsor-Investigator, Younes Oujidi, Professor Oujidi Younes, Mohammed VI University Hospital
Organization: Mohammed VI University Hospital (Other)
Other Study IDs: Critial Care
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Embolism (PE); Snake Envenomation
MeSH Terms: conditions — Pulmonary Embolism; Snake Bites

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Viper envenomation constitutes a medical emergency predominantly occurring in rural regions, where specific viper species are endemic, with their distribution influenced by climatic variations. The literature describes numerous complications associated with viper bites, including neurological disturbance, hematological abnormalities, and irreversible renal failure.

We report the case of a 65-year-old female patient admitted to the intensive care unit for viper envenomation characterized by extensive local edema. Diagnostic investigations, including laboratory tests and imaging studies, revealed the presence of a bilateral pulmonary embolism. The patient was subsequently treated with antivenom therapy, followed by initiation of low molecular weight heparin. Despite the recognized high risk of viper envenomation described in the literature, the patient experienced an uncomplicated clinical course and was discharged in stable condition with no further complications.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18years old

Exclusion Criteria:

* Not bitten by snakes

Ages: 18 Years to 100 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: People aged above 18years, developing a pulmonary embolism after snake bites
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Evolution of hematological blood test during the ICU stay | From January 2025 to May 2025

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital center Mohammed VI of Oujda, Oujda, Morocco

IPD SHARING:
Plan to Share IPD: Undecided